CLINICAL TRIAL: NCT03196284
Title: A Multi-Centre, Randomised, Open-Label, Controlled Trial Evaluating the Efficacy and Safety of Prophylactic Administration of Concizumab in Haemophilia A and B Patients With Inhibitors
Brief Title: A Trial Evaluating the Efficacy and Safety of Prophylactic Administration of Concizumab in Haemophilia A and B Patients With Inhibitors
Acronym: explorer™4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7415-4310; U1111-1179-2925 (Other: World Health Organization (WHO)); 2016-000510-30 (EudraCT Number); JapicCTI-173681 (Registry Identifier: JAPIC)
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-09

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors
MeSH Terms: interventions — concizumab; recombinant FVIIa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Concizumab (Experimental): Concizumab administered in both the main phase and extension phase, with eptacog alfa administered on-demand during bleeding episodes
  Interventions: Drug: Concizumab; Drug: Eptacog alfa
- Eptacog alfa and concizumab (Active Comparator): Eptacog alfa administered on-demand during bleeding episodes as the only intervention during the main phase. Concizumab given in the extension phase
  Interventions: Drug: Concizumab; Drug: Eptacog alfa

INTERVENTIONS:
Drug: Concizumab — A loading dose of 0.5 mg/kg will be given as the first dose, followed by 0.15 mg/kg (with potential stepwise dose escalation to 0.25 mg/kg) administered daily s.c. (subcutaneously, under the skin). Treatment duration is 24 weeks in the main trial, and up to 52 weeks in the extension phase
Drug: Eptacog alfa — A single dose of 90 μg/kg eptacog alfa one week after dosing with concizumab. On-demand treatment during bleeding episodes in both treatment arms

SUMMARY:
This trial is conducted in Africa, Asia, Europe and North America. The aim of the trial is to assess the efficacy of concizumab administered s.c. (subcutaneously, under the skin) once daily in preventing bleeding episodes in haemophilia A and B patients with inhibitors.

ELIGIBILITY:
Inclusion Criteria: - Informed consent obtained before any trial related activities. Trial related activities are any procedures that are carried out as part of the trial, including activities to determine the suitability for the trial - Male haemophilia A or B patients with inhibitors aged 18 years or older at the time of signing informed consent - Patients currently in need of treatment with bypassing agents Exclusion Criteria: - Known or suspected hypersensitivity to trial product(s) or related products - Known inherited or acquired bleeding disorder other than haemophilia - Ongoing or planned immune tolerance induction therapy or prophylaxis with FVIII or FIX

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (3):
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Iowa City, Iowa
- Novo Nordisk Investigational Site, Vienna, Austria
- Novo Nordisk Investigational Site, Toronto, Ontario, Canada
- Novo Nordisk Investigational Site, Zagreb, Croatia
- Novo Nordisk Investigational Site, Århus N, Denmark
- Novo Nordisk Investigational Site, Athens, Greece
- Novo Nordisk Investigational Site, Tel Litwinsky, Israel
- Italy (2):
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Milan
- Japan (3):
  - Novo Nordisk Investigational Site, Aichi
  - Novo Nordisk Investigational Site, Nara
  - Novo Nordisk Investigational Site, Tokyo
- Malaysia (2):
  - Novo Nordisk Investigational Site, Georgetown, Penang
  - Novo Nordisk Investigational Site, Kota Kinabalu
- Spain (2):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Seville
- Novo Nordisk Investigational Site, Solna, Sweden
- Novo Nordisk Investigational Site, Lviv, Ukraine
- United Kingdom (2):
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
According to disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Derived] Shapiro AD, Angchaisuksiri P, Astermark J, Benson G, Castaman G, Eichler H, Jimenez-Yuste V, Kavakli K, Matsushita T, Poulsen LH, Wheeler AP, Young G, Zupancic-Salek S, Oldenburg J, Chowdary P. Long-term efficacy and safety of subcutaneous concizumab prophylaxis in hemophilia A and hemophilia A/B with inhibitors. Blood Adv. 2022 Jun 14;6(11):3422-3432. doi: 10.1182/bloodadvances.2021006403. PMID 35290453
- [Derived] Shapiro AD, Angchaisuksiri P, Astermark J, Benson G, Castaman G, Chowdary P, Eichler H, Jimenez-Yuste V, Kavakli K, Matsushita T, Poulsen LH, Wheeler AP, Young G, Zupancic-Salek S, Oldenburg J. Subcutaneous concizumab prophylaxis in hemophilia A and hemophilia A/B with inhibitors: phase 2 trial results. Blood. 2019 Nov 28;134(22):1973-1982. doi: 10.1182/blood.2019001542. PMID 31444162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 17 sites in 12 countries as follows: Austria (1), Croatia (1), Denmark (1), Italy (2), Spain (2), Sweden (1), the United Kingdom (1), Israel (1), Malaysia (2), Ukraine (1), Japan (2) and the United States (2). In addition to these sites, 4 sites were approved by the IRB/IEC and/or local health authority but did not screen or assign any participants to treatment.
Pre-assignment Details: The trial consisted of two treatment periods: main part which lasted 24 weeks for participants randomised to eptacog alfa and at least 24 weeks for participants randomised to concizumab, and an extension part which lasted up to 94 weeks.
Groups:
- Concizumab- Main Part: Participants were to receive subcutaneous (s.c.) injection of concizumab once daily for 24 weeks. The initial dose was 0.15 milligrams per kilogram (mg/kg) and then the dose was escalated to 0.20 and 0.25 mg/kg based on the number of spontaneous bleeding episodes. A loading dose of 0.5 mg/kg was given as the first concizumab dose. A single injection of 90 micrograms per kilogram (μg/kg) eptacog alfa (rFVIIa) was administered in a non-bleeding state one week after the dosing with concizumab had initiated.
- Eptacog Alfa- Main Part: Participants were to receive eptacog alfa on-demand treatment for 24 weeks.
- Concizumab- Extension Part: Participants who completed main part treatment were to receive s.c. injection of concizumab once daily for 52-94 weeks. Participants who received concizumab during the main part were to continue with their treatment at last dose by the end of main part and those received eptacog alfa during the main part were to start their treatment with 0.15 mg/kg of concizumab. The dose was then escalated to 0.20 and 0.25 mg/kg based on the number of spontaneous bleeding episodes. A loading dose of 0.5 mg/kg was given as the first concizumab dose. A single injection of 90 micrograms per kilogram (μg/kg) eptacog alfa (rFVIIa) was administered in a non-bleeding state one week after dosing with concizumab had initiated.
Period: Main Part
Arm/Group | Concizumab- Main Part | Eptacog Alfa- Main Part | Concizumab- Extension Part
Started | 17 | 9 | 0
Concizumab 0.15 mg/kg (The last dose level the participants received in main part of the trial.) | 15 | 0 | 0
Concizumab 0.20 mg/kg (The last dose level the participants received in main part of the trial.) | 2 | 0 | 0
Concizumab 0.25 mg/kg (The last dose level the participants received in main part of the trial.) | 0 | 0 | 0
Completed | 17 | 8 | 0
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Extension Part
Arm/Group | Concizumab- Main Part | Eptacog Alfa- Main Part | Concizumab- Extension Part
Started | 0 (Participants who completed main part are presented in separate treatment arm.) | 0 (Participants switched to treatment with concizumab in the extension part of the study.) | 25 (Participants who completed the main part entered the extension part of the study.)
Concizumab 0.15 mg/kg (The last dose level the participants received in extension part of the trial.) | 0 | 0 | 12
Concizumab 0.20 mg/kg (The last dose level the participants received in extension part of the trial.) | 0 | 0 | 9
Concizumab 0.25 mg/kg (The last dose level the participants received in extension part of the trial.) | 0 | 0 | 4
Completed | 0 | 0 | 22
Not Completed | 0 | 0 | 3
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised participants.
Groups:
- Concizumab: Participants were to receive subcutaneous (s.c.) injection of concizumab once daily. In main part, the initial dose was 0.15 milligrams per kilogram (mg/kg) and then the dose was escalated to 0.20 and 0.25 mg/kg based on the number of spontaneous bleeding episodes. Participants who completed the main part of the study continued their treatment in the extension part for 52-94 weeks. A loading dose of 0.5 mg/kg was given as the first concizumab dose. A single injection of 90 micrograms per kilogram (μg/kg) eptacog alfa (rFVIIa) was administered in a non-bleeding state one week after dosing with concizumab had initiated.
- Eptacog Alfa: Participants were to receive eptacog alfa on-demand treatment for 24 weeks in main part. All participants were then switched to concizumab treatment in the extension part.
- Total: Total of all reporting groups
Arm/Group | Concizumab | Eptacog Alfa | Total
Number analyzed (Participants) | 17 | 9 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.1 (11.1) | 41.1 (15.0) | 36.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17 | 9 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 16 | 9 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 5 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number of Bleeding Episodes
Description: The number of bleeding episodes that were treated during at least 24 weeks from treatment onset (week 0) are presented.
Time Frame: During at least 24 weeks from treatment onset (week 0)
Population: The FAS included all randomised participants.
Measure: Number; unit: episodes
Groups:
- Concizumab- Main Part: Participants were to receive s.c. injection of concizumab once daily for 24 weeks. The initial dose was 0.15 mg/kg and then the dose was escalated to 0.20 and 0.25 mg/kg based on the number of spontaneous bleeding episodes. A loading dose of 0.5 mg/kg was given as the first concizumab dose. A single injection of 90 micrograms per kilogram (μg/kg) eptacog alfa (rFVIIa) was administered in a non-bleeding state one week after the dosing with concizumab had initiated.
Arm/Group | Concizumab- Main Part | Eptacog Alfa- Main Part
Number analyzed (Participants) | 17 | 9
episodes | 47 | 77

2. Secondary Outcome: The Number of Bleeding Episodes
Description: The number of bleeding episodes that were treated during at least 76 weeks from treatment onset (week 0) are presented. This outcome measure is applicable for only 'Concizumab' treatment arm.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: The FAS included all randomised participants.
Measure: Number; unit: episodes
Groups:
- Concizumab: Participants were to receive s.c. injection of concizumab once daily. In main part, the initial dose was 0.15 mg/kg and then the dose was escalated to 0.20 and 0.25 mg/kg based on the number of spontaneous bleeding episodes. Participants who completed the main part of the study continued their treatment in the extension part for 52-94 weeks. A loading dose of 0.5 mg/kg was given as the first concizumab dose. A single injection of 90 μg/kg eptacog alfa (rFVIIa) was administered in a non-bleeding state one week after dosing with concizumab had initiated.
Arm/Group | Concizumab
Number analyzed (Participants) | 25
episodes | 256

3. Secondary Outcome: The Number of Spontaneous Bleeding Episodes
Description: Bleeds that were not linked to a specific, known action or event are called spontaneous bleeding episodes. The number of spontaneous bleeding episodes that were treated during at least 24 weeks from treatment onset (week 0) are presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 24 weeks from treatment onset (week 0)
Population: The FAS included all randomised participants.
Measure: Number; unit: episodes
Groups:
- Concizumab 0.15 mg/kg- Main Part: Participants received s.c. injection of 0.15 mg/kg concizumab once daily for 24 weeks. A loading dose of 0.5 mg/kg was given as the first concizumab dose.
- Concizumab 0.20 mg/kg- Main Part: Participants received s.c. injection of concizumab once daily for 24 weeks. The initial dose was 0.15 mg/kg which was then escalated to 0.20 mg/kg based on the number of spontaneous bleeding episodes. A loading dose of 0.5 mg/kg was given as the first concizumab dose.
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Eptacog Alfa- Main Part
Number analyzed (Participants) | 15 | 2 | 9
episodes | 19 | 5 | 69

4. Secondary Outcome: The Number of Spontaneous Bleeding Episodes
Description: Bleeds that were not linked to a specific, known action or event are called spontaneous bleeding episodes. The number of spontaneous bleeding episodes that were treated during at least 76 weeks from treatment onset (week 0) are presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: The FAS included all randomised participants.
Measure: Number; unit: episodes
Groups:
- Concizumab 0.15 mg/kg: Participants were to receive s.c. injection of 0.15 mg/kg of concizumab once daily. Participants who completed the main part (24 weeks) of the study continued their treatment in the extension part for 52-94 weeks. Participants who received concizumab during the main part were to continue with their treatment at last dose by the end of main part and those received eptacog alfa during the main part were to start their treatment with concizumab. A loading dose of 0.5 mg/kg was given as the first concizumab dose. A single injection of 90 μg/kg eptacog alfa (rFVIIa) was administered in a non-bleeding state one week after dosing with concizumab had initiated.
- Concizumab 0.20 mg/kg: Participants were to receive s.c. injection of concizumab once daily. Participants who completed the main part (24 weeks) of the study continued their treatment in the extension part for 52-94 weeks. Participants who received concizumab during the main part were to continue with their treatment at last dose by the end of main part and those received eptacog alfa during the main part were to start their treatment with concizumab. The initial dose was 0.15 mg/kg which was then escalated to 0.20 mg/kg based on the number of spontaneous bleeding episodes. A loading dose of 0.5 mg/kg was given as the first concizumab dose. A single injection of 90 μg/kg eptacog alfa (rFVIIa) was administered in a non-bleeding state one week after dosing with concizumab had initiated.
- Concizumab 0.25 mg/kg: Participants were to receive s.c. injection of concizumab once daily. Participants who completed the main part (24 weeks) of the study continued their treatment in the extension part for 52-94 weeks. Participants who received concizumab during the main part were to continue with their treatment at last dose by the end of main part and those received eptacog alfa during the main part were to start their treatment with concizumab. The initial dose was 0.15 mg/kg which was then escalated to 0.25 mg/kg based on the number of spontaneous bleeding episodes. A loading dose of 0.5 mg/kg was given as the first concizumab dose. A single injection of 90 μg/kg eptacog alfa (rFVIIa) was administered in a non-bleeding state one week after dosing with concizumab had initiated.
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 12 | 9 | 4
episodes | 36 | 9 | 7

5. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) During at Least 24 Weeks From Treatment Onset
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a medicinal product, and which does not necessarily had a causal relationship with this treatment. A TEAE was defined as an event that had onset from the first exposure to treatment until the last visit in the trial. Number of TEAEs that occurred during at least 24 weeks from treatment onset (week 0) are presented. The data is presented per the dose level which the participants have reached at the time of event.
Time Frame: During at least 24 weeks from treatment onset (week 0)
Population: The safety analysis set (SAS) included all randomised participants.
Measure: Number; unit: events
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Eptacog Alfa- Main Part
Number analyzed (Participants) | 17 | 2 | 9
events | 39 | 4 | 18

6. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) During at Least 76 Weeks From Treatment Onset
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a medicinal product, and which does not necessarily had a causal relationship with this treatment. A TEAE was defined as an event that had onset from the first exposure to treatment until the last visit in the trial. Number of TEAEs that occurred during at least 76 weeks from treatment onset (week 0) are presented. The data is presented per the dose level which the participants have reached at the time of event.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: The SAS included all randomised participants. Overall number of participants analysed = number of participants contributed to the analysis at the particular dose level.
Measure: Number; unit: events
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 25 | 13 | 4
events | 104 | 24 | 3

7. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) Within 24 Hours After Eptacog Alfa Administration
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a medicinal product, and which does not necessarily had a causal relationship with this treatment. A TEAE was defined as an event that had onset from the first exposure to treatment until the last visit in the trial. Number of TEAEs that occurred within 24 hours after eptacog alfa administration are presented. This outcome measure is applicable only for 'Eptacog alfa' treatment arm.
Time Frame: Within 24 hours after eptacog alfa administration
Population: The SAS included all randomised participants.
Measure: Number; unit: events
Arm/Group | Eptacog Alfa- Main Part
Number analyzed (Participants) | 9
events | 0

8. Secondary Outcome: Occurrence of Anti-concizumab Antibodies During at Least 24 Weeks From Treatment Onset
Description: Occurrence of anti-concizumab antibodies during at least 24 weeks from treatment onset (week 0) is presented. This outcome measure is applicable for only 'Concizumab' treatment arm.
Time Frame: During at least 24 weeks from treatment onset (week 0)
Population: The FAS included all participants who received concizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Concizumab- Main Part
Number analyzed (Participants) | 17
Participants
  Yes | 3
  No | 14

9. Secondary Outcome: Occurrence of Anti-concizumab Antibodies During at Least 76 Weeks From Treatment Onset
Description: Occurrence of anti-concizumab antibodies during at least 76 weeks from treatment onset (week 0) is presented. This outcome measure is applicable for only 'Concizumab' treatment arm.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: The FAS included all participants who received concizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Concizumab
Number analyzed (Participants) | 25
Participants
  Yes | 6
  No | 19

10. Secondary Outcome: Change in Fibrinogen
Description: Change in fibrinogen during at least 24 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 24 weeks from treatment onset (week 0)
Population: The SAS included all randomised participants. Overall number of participants analysed = number of participants available for analysis.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Eptacog Alfa- Main Part
Number analyzed (Participants) | 14 | 2 | 8
Grams per liter (g/L) | -0.24 (0.45) | -1.24 (1.61) | 0.13 (0.48)

11. Secondary Outcome: Change in Fibrinogen
Description: Change in fibrinogen during at least 76 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: The SAS included all randomised participants. Overall number of participants analysed = number of participants available for the analysis.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 11 | 9 | 3
g/L | -0.14 (0.51) | -0.56 (0.72) | -1.51 (1.44)

12. Secondary Outcome: Change in D-dimer
Description: Change in D-dimer during at least 24 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 24 weeks from treatment onset (week 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Eptacog Alfa- Main Part
Number analyzed (Participants) | 15 | 2 | 8
Nanograms per milliliter (ng/mL) | 227 (239) | 550 (608) | -48 (614)

13. Secondary Outcome: Change in D-dimer
Description: Change in D-dimer during at least 76 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 11 | 9 | 3
ng/mL | 308 (601) | 193 (912) | 340 (887)

14. Secondary Outcome: Change in Prothrombin Fragment 1 + 2 (F1 + 2)
Description: Change in F1 + 2 during at least 24 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 24 weeks from treatment onset (week 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Picomoles per liter (pmol/L)
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Eptacog Alfa- Main Part
Number analyzed (Participants) | 15 | 2 | 8
Picomoles per liter (pmol/L) | 154 (256) | 164 (1) | 0 (33)

15. Secondary Outcome: Change in Prothrombin Fragment 1 + 2 (F1 + 2)
Description: Change in F1 + 2 during at least 76 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 11 | 9 | 3
pmol/L | 159 (202) | 457 (458) | 349 (452)

16. Secondary Outcome: Change in Prothrombin Time (PT)
Description: Change in PT during at least 24 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 24 weeks from treatment onset (week 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Seconds (sec)
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Eptacog Alfa- Main Part
Number analyzed (Participants) | 15 | 2 | 7
Seconds (sec) | 0.2 (0.4) | -1.0 (1.0) | 0.0 (0.5)

17. Secondary Outcome: Change in Prothrombin Time (PT)
Description: Change in PT during at least 76 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 11 | 9 | 3
sec | -0.4 (0.6) | 0.4 (0.6) | 0.3 (0.5)

18. Secondary Outcome: Change in Activated Partial Thromboplastin Time (APTT)
Description: Change in APTT during at least 24 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 24 weeks from treatment onset (week 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Eptacog Alfa- Main Part
Number analyzed (Participants) | 15 | 2 | 7
sec | -2.6 (12.1) | 0.9 (2.3) | 5.9 (15.2)

19. Secondary Outcome: Change in Activated Partial Thromboplastin Time (APTT)
Description: Change in APTT during at least 76 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 11 | 9 | 3
sec | -6.6 (9.0) | 3.7 (6.9) | 20.9 (17.3)

20. Secondary Outcome: Change in Anti-thrombin (AT)
Description: Change in AT during at least 24 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 24 weeks from treatment onset (week 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage point of AT
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Eptacog Alfa- Main Part
Number analyzed (Participants) | 15 | 2 | 8
Percentage point of AT | -1 (11) | 8 (4) | 1 (10)

21. Secondary Outcome: Change in Anti-thrombin (AT)
Description: Change in AT after at least 76 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: After at least 76 weeks from treatment onset (week 0)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percentage point of AT
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 11 | 9 | 3
Percentage point of AT | -3 (15) | -5 (11) | -1 (14)

22. Secondary Outcome: Concentration of Concizumab
Description: Concentration of concizumab prior to the last dose administration at 24 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration at 24 weeks
Population: The FAS included all randomised participants.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part
Number analyzed (Participants) | 15 | 2
ng/mL | 350.6 (316.8) | 517.5 (309.0)

23. Secondary Outcome: Concentration of Concizumab
Description: Concentration of concizumab prior to the last dose administration after atleast 76 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration after atleast 76 weeks
Population: The FAS included all randomised participants. Overall number of participants analysed = number of participants available for the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 11 | 9 | 3
ng/mL | 205.5 (254.5) | 1354.7 (1004.3) | 941.7 (943.1)

24. Secondary Outcome: Free Tissue Factor Pathway Inhibitor (TFPI) Concentration Value
Description: Free TFPI (TFPI not bound to concizumab) concentration value prior to the last dose administration at 24 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration at 24 weeks
Population: The FAS included all randomised participants. Overall number of participants analysed = number of participants available for analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Eptacog Alfa- Main Part
Number analyzed (Participants) | 15 | 2 | 8
ng/mL | 29.9 (9.6) | 4.8 (0.0) | 94.3 (13.8)

25. Secondary Outcome: Free Tissue Factor Pathway Inhibitor (TFPI) Concentration Value
Description: Free TFPI concentration value prior to the last dose administration after atleast 76 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration after atleast 76 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 11 | 9 | 3
ng/mL | 30.3 (28.2) | 8.3 (4.9) | 12.2 (12.9)

26. Secondary Outcome: Peak Thrombin Generation
Description: Peak thrombin generation is the maximal concentration of thrombin formed at a given point in time. Peak thrombin generation prior to the last dose administration at 24 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration at 24 weeks
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Nanomoles per liter (nmol/L)
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Eptacog Alfa- Main Part
Number analyzed (Participants) | 15 | 2 | 1
Nanomoles per liter (nmol/L) | 57.8 (28.9) | 119.0 (12.7) | 12.0 (NA) — Standard deviation could not be calculated as only 1 participant was available for analysis.

27. Secondary Outcome: Peak Thrombin Generation
Description: Peak thrombin generation is the maximal concentration of thrombin formed at a given point in time. Peak thrombin generation prior to the last dose administration after atleast 76 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration after atleast 76 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 11 | 9 | 3
nmol/L | 79.5 (55.3) | 98.7 (20.4) | 75.7 (30.6)

28. Secondary Outcome: Endogenous Thrombin Potential
Description: Endogenous thrombin potential prior to the last dose administration at 24 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration at 24 weeks
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Nanomolar*minute (nM*min)
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Eptacog Alfa- Main Part
Number analyzed (Participants) | 15 | 2 | 1
Nanomolar*minute (nM*min) | 901.5 (347.6) | 1589.5 (133.6) | 228.0 (NA) — Standard deviation could not be calculated as only 1 participant was available for analysis.

29. Secondary Outcome: Endogenous Thrombin Potential
Description: Endogenous thrombin potential prior to the last dose administration after at least 76 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration after atleast 76 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: nM*min
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 11 | 9 | 3
nM*min | 1056.5 (438.5) | 1356.9 (223.9) | 1178.0 (184.3)

30. Secondary Outcome: Thrombin Generation Velocity Index
Description: Thrombin generation velocity index prior to the last dose administration at 24 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration at 24 weeks
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: nM/min
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Eptacog Alfa- Main Part
Number analyzed (Participants) | 15 | 2 | 1
nM/min | 5.3 (3.3) | 14.5 (3.5) | 1.0 (NA) — Standard deviation could not be calculated as only 1 participant was available for analysis.

31. Secondary Outcome: Thrombin Generation Velocity Index
Description: Thrombin generation velocity index prior to the last dose administration after at least 76 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration after atleast 76 weeks
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: nM/min
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 11 | 9 | 3
nM/min | 10.0 (12.0) | 9.7 (3.5) | 6.7 (3.2)

ADVERSE EVENTS:
Time Frame: From start of study drug administration (week 0) up to 126 weeks
Description: Results are based on the safety analysis set which included all randomized participants.
  All presented adverse events are treatment emergent adverse events (TEAEs). TEAE was defined as an event that had onset from the first exposure to treatment (randomisation date, in case of on-demand arm) until the last visit in the trial.
Groups:
- Concizumab 0.15 mg/kg- Extension Part: Participants who were on treatment with concizumab once daily at the end of main part of the study continued their treatment in the extension part. Participants who received eptacog alfa in the main part switched to treatment with concizumab in the extension part (a loading dose of 0.5 mg/kg was given as the first concizumab dose). The dose of concizumab was 0.15 mg/kg.
- Concizumab 0.20 mg/kg- Extension Part: Participants who were on treatment with concizumab once daily at the end of main part of the study continued their treatment in the extension part. Participants who received eptacog alfa in the main part switched to treatment with concizumab in the extension part (a loading dose of 0.5 mg/kg was given as the first concizumab dose). The initial dose of concizumab was 0.15 mg/kg which was then escalated to 0.20 mg/kg based on the number of spontaneous bleeding episodes.
- Concizumab 0.25 mg/kg- Extension Part: Participants who were on treatment with concizumab once daily at the end of main part of the study continued their treatment in the extension part. Participants who received eptacog alfa in the main part switched to treatment with concizumab in the extension part (a loading dose of 0.5 mg/kg was given as the first concizumab dose). The initial dose of concizumab was 0.15 mg/kg which was then escalated to 0.25 mg/kg based on the number of spontaneous bleeding episodes.
Arm/Group | Eptacog Alfa- Main Part | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Concizumab 0.15 mg/kg- Extension Part | Concizumab 0.20 mg/kg- Extension Part | Concizumab 0.25 mg/kg- Extension Part
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/17 | 0/2 | 0/23 | 0/13 | 0/4
Serious Adverse Events (participants affected / at risk) | 3/9 | 1/17 | 0/2 | 3/23 | 1/13 | 0/4
Other Adverse Events (participants affected / at risk) | 7/9 | 13/17 | 2/2 | 13/23 | 9/13 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eptacog Alfa- Main Part (N=9) | Concizumab 0.15 mg/kg- Main Part (N=17) | Concizumab 0.20 mg/kg- Main Part (N=2) | Concizumab 0.15 mg/kg- Extension Part (N=23) | Concizumab 0.20 mg/kg- Extension Part (N=13) | Concizumab 0.25 mg/kg- Extension Part (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central venous catheter removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eptacog Alfa- Main Part (N=9) | Concizumab 0.15 mg/kg- Main Part (N=17) | Concizumab 0.20 mg/kg- Main Part (N=2) | Concizumab 0.15 mg/kg- Extension Part (N=23) | Concizumab 0.20 mg/kg- Extension Part (N=13) | Concizumab 0.25 mg/kg- Extension Part (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 3 (6) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prothrombin fragment 1.2 increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prothrombin level increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulnar nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 3 (5) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT03196284/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT03196284/SAP_001.pdf